CLINICAL TRIAL: NCT05569096
Title: Clinical Significance of Circulating T Regulatory Cells , Soluble CD25 and CXCL9 to Assess Disease Activity of Vitiligo.
Brief Title: Tregs CD25 CXCL9 in Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jian Hashim Mohammed , MD, Assistant Lecturer, Assiut University
Other Study IDs: Tregs CD25 CXCL9 vitiligo
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Vitiligo; CD25 Deficiency; Chemokine (C-X-C Motif); Tregs
MeSH Terms: conditions — Vitiligo; Interleukin 2 Receptor, Alpha, Deficiency of

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ELIZA , Flowcytometry — CD25 , CXCL9 by ELISA. T cell population , T regulatory cells by Flow cytometry.

SUMMARY:
Clinical significance of circulating T regulatory cells , soluble CD25 and CXCL9 to assess disease activity of vitiligo.

DETAILED DESCRIPTION:
Vitiligo is an acquired and polygenic skin depigmenting disease characterized by bilateral, symmetrical depigmented patches over the entire body.

Its pathogenesis is multifactorial; however, the exact mechanisms that integrate the individual genetic susceptibility, melanocyte auto aggression, and failure of immune tolerance mechanisms are still not fully understood. The presence of these autoreactive CD8+ and CD4+ T cells in vitiligo patients' skin and blood samples . indicates a dysregulation of regulatory T-cell mechanism, which can suppress these cells.

Previous studies have reported an altered Treg cell frequency and function in vitiligo patients.

FoxP3 is the key transcriptional regulators of Tregs which mediate Treg cell function by repressing the expression of cytokines (IL2 and IL4 ) and upregulate the Treg cell markers (CTLA-4 and CD25 ).

Expression of IL-2 and its receptor CD25 are the most fundamental events in the host immune response. Thus any disorder in which T lymphocyte activation occurs at a substantial level is expected to induce expression of CD25 beyond ambient levels; this had been reported in atopic asthma, multiple sclerosis, allergic responses.

CD4+ CD25 FoxP3+ Tregs are important in maintaining self-tolerance and regulating immune responses in both physiological and pathological conditions .

Chemokines are important inflammatory factors that participate in many autoimmune responses.

C-X-C motif chemokine ligand 9 (CXCL9) is linked to the Th1 pattern and has been suggested as one of the most relevant chemokine axes that promote T-cell migration in different autoimmune and inflammatory processes.

In vitiligo, CXCL9 has been suggested to promote melanocyte-specic CTLs to in ltrate into the basal layer of the epidermis to attack melanocytes, resulting in the deficiency of melanin.

ELIGIBILITY:
Inclusion Criteria:The patients will be enrolled in the study if they have :-

* Non segmental vitiligo.

Exclusion Criteria:

The following patients were excluded from this study:

* Patients receiving systemic treatment in the last two months.
* Patients with any autoimmune disease, such as rheumatoid arthritis. inflammatory bowel disease, psoriasis, or systemic lupus erythematosus; patients with type 1 diabetes mellitus.
* Patients with any thyroid and/or neoplastic diseases.

Ages: 15 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study include 50 patients with clinically diagnosed vitiligo. Eligible patients are those attending the dermatology, venereology, and andrology outpatient clinic at Assiut University Hospital.
  Separately, the control group included 40 healthy subjects who were matched to vitiligo patients according to age and sex.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To assess role of circulating T regulatory cells, soluble CD25 and CXCL9 in disease activity of vitiligo | Baseline
  compare presences of T regulatory cells , soluble CD25 and CXCL9 between healthy control and vitiligo patients.
  To assess role of circulating T regulatory cells, soluble CD25 and CXCL9 in disease activity of vitiligo

REFERENCES:
- [Background] Gharib K, Gadallah H, Elsayed A. Chemokines in Vitiligo Pathogenesis: CXCL10 and 12. J Clin Aesthet Dermatol. 2021 Sep;14(9):27-32. PMID 34980968
- [Background] Marchioro HZ, Silva de Castro CC, Fava VM, Sakiyama PH, Dellatorre G, Miot HA. Update on the pathogenesis of vitiligo. An Bras Dermatol. 2022 Jul-Aug;97(4):478-490. doi: 10.1016/j.abd.2021.09.008. Epub 2022 May 25. PMID 35643735
- [Background] Bergqvist C, Ezzedine K. Vitiligo: A Review. Dermatology. 2020;236(6):571-592. doi: 10.1159/000506103. Epub 2020 Mar 10. PMID 32155629
- [Background] Giri PS, Dwivedi M, Laddha NC, Begum R, Bharti AH. Altered expression of nuclear factor of activated T cells, forkhead box P3, and immune-suppressive genes in regulatory T cells of generalized vitiligo patients. Pigment Cell Melanoma Res. 2020 Jul;33(4):566-578. doi: 10.1111/pcmr.12862. Epub 2020 Jan 23. PMID 31917889
- [Background] Yang L, Yang S, Lei J, Hu W, Chen R, Lin F, Xu AE. Role of chemokines and the corresponding receptors in vitiligo: A pilot study. J Dermatol. 2018 Jan;45(1):31-38. doi: 10.1111/1346-8138.14004. Epub 2017 Nov 8. PMID 29115683
- [Background] Yang L, Wei Y, Sun Y, Shi W, Yang J, Zhu L, Li M. Interferon-gamma Inhibits Melanogenesis and Induces Apoptosis in Melanocytes: A Pivotal Role of CD8+ Cytotoxic T Lymphocytes in Vitiligo. Acta Derm Venereol. 2015 Jul;95(6):664-70. doi: 10.2340/00015555-2080. PMID 25721262